CLINICAL TRIAL: NCT07150312
Title: Can Different Exercise Modalities Improve Esports Performance? Study Protocol for a 12-week Three-arm Randomized Controlled Trial
Brief Title: Can Different Exercise Modalities Improve Esports Performance?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ma Ruisi (Other)
Responsible Party: Sponsor-Investigator, Ma Ruisi, Co-Investigator, Jinan University Guangzhou
Organization: Jinan University Guangzhou (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SBRE-24-0942
Record Dates: First submitted 2025-08-17; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Esports Players

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-intensity interval training (HIIT) group (Experimental): A 12-week home-based HIIT exercise plan (running). Duration: Each session consists of 10 x 1-minute high-intensity bouts interspersed with 10 x 1-minute recovery periods. Adding the 3-minute warmup and 3-minute cool-down, each session totals approximately 26 minutes. This protocol is followed for 12 weeks.
  Intensity: High-intensity bouts are performed at 80-90% of HRmax (RPE 15-18). Recovery periods are at 40-50% of HRmax (RPE 11-13). Warm-up and cool-down are at 50% HRmax (RPE 11-13).
  Modality: Running, jogging, or brisk walking, either on a treadmill or outdoors.
  Supervision: The first three sessions are supervised in a laboratory setting. Subsequent sessions are unsupervised and performed at home with heart rate monitoring and remote data tracking via Polar Flow for Coach.
  Interventions: Behavioral: HIIT
- Moderate-intensity continuous training (MICT) group (Experimental): A 12-week home-based MICT exercise plan (running). Duration: Each session consists of 20 minutes of continuous exercise. Including the 3-minute warm-up and 3-minute cool-down, each session totals 26 minutes. This protocol is followed for 12 weeks.
  Intensity: Exercise is performed at 64-76% of HRmax (RPE 12-14). Warm-up and cool-down are at 50% HRmax (RPE 11-13).
  Modality: Running, jogging, or brisk walking, either on a treadmill or outdoors.
  Supervision: The first three sessions are supervised in a laboratory setting. Subsequent sessions are unsupervised and performed at home with heart rate monitoring and remote data tracking via Polar Flow for Coach.
  Interventions: Behavioral: MICT
- Control (No Intervention): No intervention. Members of the control group are required to maintain their usual habits of gaming, sleeping, eating, and exercising. The experiment does not implement any interventions for the control group.

INTERVENTIONS:
Behavioral: HIIT — A 12-week home-based HIIT exercise plan (running). Duration: Each session consists of 10 x 1-minute high-intensity bouts interspersed with 10 x 1-minute recovery periods. Adding the 3-minute warmup and 3-minute cool-down, each session totals approximately 26 minutes. This protocol is followed for 12 weeks.
  Intensity: High-intensity bouts are performed at 80-90% of HRmax (RPE 15-18). Recovery periods are at 40-50% of HRmax (RPE 11-13). Warm-up and cool-down are at 50% HRmax (RPE 11-13).
  Modality: Running, jogging, or brisk walking, either on a treadmill or outdoors.
  Supervision: The first three sessions are supervised in a laboratory setting. Subsequent sessions are unsupervised and performed at home with heart rate monitoring and remote data tracking via Polar Flow for Coach.
  Arms: High-intensity interval training (HIIT) group
Behavioral: MICT — A 12-week home-based MICT exercise plan (running). Duration: Each session consists of 20 minutes of continuous exercise. Including the 3-minute warm-up and 3-minute cool-down, each session totals 26 minutes. This protocol is followed for 12 weeks.
  Intensity: Exercise is performed at 64-76% of HRmax (RPE 12-14). Warm-up and cool-down are at 50% HRmax (RPE 11-13).
  Modality: Running, jogging, or brisk walking, either on a treadmill or outdoors.
  Supervision: The first three sessions are supervised in a laboratory setting. Subsequent sessions are unsupervised and performed at home with heart rate monitoring and remote data tracking via Polar Flow for Coach.
  Arms: Moderate-intensity continuous training (MICT) group

SUMMARY:
This study aims to investigate the long-term effects of high-intensity interval training (HIIT) and moderate-intensity continuous training (MICT) on esports performance through a 12-week three-arm randomized controlled trial, and to examine the sustainability of these effects during a follow-up period after intervention cessation. Additionally, we seek to compare the differential impacts of these two exercise modalities on various dimensions of esports performance, thereby providing evidence-based guidance for esports training regimens and enhancing our understanding of the underlying mechanisms by which different exercise approaches influence cognitive and motor capabilities essential for competitive gaming.

ELIGIBILITY:
Inclusion Criteria:

1. 18-29 years old;
2. regular FPS players engaging in shooters within the past six months;
3. healthy individuals who are capable of physical tests or HIIT;
4. no regular exercise habits;
5. can understand English or Chinese.

Exclusion Criteria:

1. self-reported history of neurological, psychiatric, or medical diseases;
2. current intake of medications and/or recreational drugs that could affect the central nervous system and/or the ability to learn;
3. not a regular user of Aim Lab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Esports performance | Baseline (pre-intervention) and immediately after 12-week intervention completion
  Measured by Aim Lab (Online shooting program) and esports-related mental quality questionnaire.

OTHER OUTCOMES:
VO2max | Baseline (pre-intervention) and immediately after 12-week intervention completion
  Progressive Aerobic Cardiovascular Endurance Run 20-m (measured in laps)
Handgrip | Baseline (pre-intervention) and immediately after 12-week intervention completion
  Handgrip dynamometer (measured in kilograms)
Core strength | Baseline (pre-intervention) and immediately after 12-week intervention completion
  Plank test (measured in second)
Balance | Baseline (pre-intervention) and immediately after 12-week intervention completion
  Unipedal stance test (measured in second)
Agility | Baseline (pre-intervention) and immediately after 12-week intervention completion
  Agility T-test (measured in second)
Flexibility | Baseline (pre-intervention) and immediately after 12-week intervention completion
  Sit and Reach Test
Body composition (measured in centimeter) | Baseline (pre-intervention) and immediately after 12-week intervention completion
  Bioelectrical impedance analysis (BIA) device (MC-780MA)
Physical Activity Level | Baseline (pre-intervention) and immediately after 12-week intervention completion
  International Physical Activity Questionnaire (IPAQ) long form (measured in MET-minutes/week, range: 0 to no upper limit, with higher scores indicating higher levels of physical activity)
Sleep Quality | Baseline (pre-intervention) and immediately after 12-week intervention completion
  Pittsburgh Sleep Quality Index (PSQI) (scored from 0 to 21, with higher scores indicating worse sleep quality)
Total Energy Intake | Baseline (pre-intervention) and immediately after 12-week intervention completion
  Daily caloric intake measured by a validated 3-day food diary (measured in kilocalories/day)
Carbohydrate Intake | Baseline (pre-intervention) and immediately after 12-week intervention completion
  Daily carbohydrate consumption measured by validated 3-day food diary (measured in grams/day)
Fat Intake | Baseline (pre-intervention) and immediately after 12-week intervention completion
  Daily fat consumption measured by a validated 3-day food diary (measured in grams/day)
Protein Intake | Baseline (pre-intervention) and immediately after 12-week intervention completion
  Daily protein consumption measured by a validated 3-day food diary (measured in grams/day)
Affect | Baseline (pre-intervention) and immediately after 12-week intervention completion
  Positive and Negative Affect Schedule (PANAS), a 20-item scale measuring both positive affect (10 items) and negative affect (10 items).Two separate scores calculated: positive affect score (range: 10-50, higher scores indicate higher positive affect) and negative affect score (range: 10-50, higher scores indicate higher negative affect)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DE Las Heras B, Li O, Rodrigues L, Nepveu JF, Roig M. Exercise Improves Video Game Performance: A Win-Win Situation. Med Sci Sports Exerc. 2020 Jul;52(7):1595-1602. doi: 10.1249/MSS.0000000000002277. PMID 31977638